CLINICAL TRIAL: NCT02175433
Title: A Phase 1 Study Evaluating Safety, Tolerability, and Pharmacokinetics of Escalating Doses of AGS67E Given as Monotherapy in Subjects With Refractory or Relapsed Lymphoid Malignancies
Brief Title: A Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Escalating Doses of AGS67E Given as Monotherapy in Subjects With Refractory or Relapsed Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AGS67E-14-1
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Relapsed Lymphoid Malignancy; Refractory Lymphoid Malignancy
Keywords: Refractory or relapsed chronic lymphocytic leukemia (CLL) prolymphocytic leukemia (PLL); Relapsed lymphoid malignancy; Refractory lymphoid malignancy; Pharmacokinetics of AGS67E; hairy cell leukemia (HCL); AGS67C; non-Hodgkin lymphoma (NHL); AGS67E
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Leukemia, Hairy Cell; Lymphoma, Non-Hodgkin | interventions — AGS67E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Dose Escalation of AGS67E 0.05 mg/kg Without GF (Experimental): Participants will receive 0.05 milligram per kilogram (mg/kg) AGS67E without growth factor (GF) by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Escalation of AGS67E 0.1 mg/kg Without GF (Experimental): Participants will receive 0.1 mg/kg AGS67E without GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Escalation of AGS67E 0.3 mg/kg Without GF (Experimental): Participants will receive 0.3 mg/kg AGS67E without GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Escalation of AGS67E 0.6 mg/kg Without GF (Experimental): Participants will receive 0.6 mg/kg AGS67E without GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Escalation of AGS67E 0.9 mg/kg Without GF (Experimental): Participants will receive 0.9 mg/kg AGS67E without GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Escalation of AGS67E 1.2 mg/kg Without GF (Experimental): Participants will receive 1.2 mg/kg AGS67E without GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Expansion of AGS67E 0.9 mg/kg Without GF (Experimental): Participants will receive 0.9 mg/kg AGS67E without GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Escalation of AGS67E 1.2 mg/kg With GF (Experimental): Participants will receive 1.2 mg/kg AGS67E with GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Escalation of AGS67E 1.5 mg/kg With GF (Experimental): Participants will receive 1.5 mg/kg AGS67E with GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Escalation of AGS67E 1.8 mg/kg With GF (Experimental): Participants will receive 1.8 mg/kg AGS67E with GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- Dose Expansion of AGS67E 1.5 mg/kg With GF (Experimental): Participants will receive 1.5 mg/kg AGS67E with GF by intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E

INTERVENTIONS:
Drug: AGS67E — intravenous (IV) infusion

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of AGS67E both without and with myeloid growth factor (GF) in subjects with refractory or relapsed lymphoid malignancies. Immunogenicity and anticancer activity of AGS67E will also be assessed.

DETAILED DESCRIPTION:
The dose escalation study will have two parts:

1. Dose Escalation of AGS67E without myeloid growth factor (GF)
2. Dose Escalation of AGS67E with myeloid growth factor (GF)

Subjects will be enrolled sequentially into dose cohorts starting with AGS67E without GF.

All subjects will receive a single 30 minute intravenous (IV) infusion of AGS67E once every three weeks. Subjects will continue treatment until disease progression, intolerability of AGS67E, investigator decision or consent withdrawal.

This dose escalation will first determine the maximum tolerated dose (MTD) of AGS67E without GF and then determine the MTD of AGS67E with GF. Once an MTD has been established, the study may enroll subjects into respective expansion cohorts of 12 subjects each at doses recommended by the data review team (DRT) (expansion cohort without GF and/or expansion cohort with GF).

During dose escalation, the Data Review Team will review cumulative unaudited data on an interim basis to review subject safety, recommend exploring additional doses and/or schedules, or the expansion of existing cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or relapsed chronic lymphocytic leukemia (CLL), prolymphocytic leukemia (PLL), hairy cell leukemia (HCL) or non-Hodgkin lymphoma (NHL) (including those of T cell origin)
* Eastern Cooperative Oncology Group performance score (ECOG) ≤ 2
* Negative pregnancy test (women of childbearing potential)
* Hematologic function, as follows (no platelet transfusion within 2 weeks and no RBC transfusion within 4 days before the first dose of study drug)

  * Absolute neutrophil count (ANC) ≥ 1,000/μL
  * Platelets ≥ 75,000/μL
  * Hemoglobin ≥ 8 g/dL (may be transfused ≥ 5 days)
* Renal function: serum creatinine ≤ 2.0 mg/dL and estimated creatinine clearance of ≥ 45 mL/min by the Cockcroft-Gault equation
* Direct bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Serum albumin ≥ 2.5 g/dL
* Aspartate aminotransferase (AST) ≤ 1.5 x ULN unless there is hepatic involvement, then 3 x ULN
* Alanine aminotransferase (ALT) ≤ 1.5 x ULN unless there is hepatic involvement, then 3 x ULN
* Sexually active fertile subjects, and their partners, must agree to use medically accepted double-barrier methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the study and at least 6 weeks after termination of study therapy

Exclusion Criteria:

* Preexisting sensory and/or motor neuropathy Grade ≥ 2
* Small molecule therapy, radiotherapy, immunotherapy, monoclonal antibodies, or chemotherapy within 2 weeks before first dose of study drug
* Radioimmunotherapy within 4 weeks before first dose of study drug
* Use of any investigational drug (including marketed drugs not approved for this indication) within 14 days prior to the first dose of study drug
* Any P-gp inducers/inhibitors or strong CYP3A inhibitors within 2 weeks before the first dose of study drug (See Appendix F for list of excluded drugs)
* Anti Graft-Versus-Host Disease (GVHD) therapy within 12 weeks before the first dose of study drug
* Platelet transfusion within 2 weeks and RBC transfusion within 4 days before the first dose of study drug
* Known central nervous system (CNS) disease
* History of other primary malignancy (including myeloid malignancy, e.g., myelodysplastic syndrome), unless

  * Curatively resected nonmelanomatous skin cancer
  * Other malignancy curatively treated with no known active disease present and no systemic treatment administered for 3 years before the first dose of study drug
* Active angina or Class III or IV Congestive Heart Failure (CHF) (New York Heart Association CHF Functional Classification System) or clinically significant cardiac disease within 12 months of the first dose of study drug, including myocardial infarction, unstable angina, Grade 2 or greater peripheral vascular disease, congestive heart failure, uncontrolled hypertension, or arrhythmias not controlled by outpatient medication
* Women who are pregnant or lactating
* Known HIV positive or AIDS
* Positive Hepatitis B surface antigen test
* Decompensated liver disease as evidenced by clinically significant ascites refractory to diuretic therapy, hepatic encephalopathy, or coagulopathy
* Known sensitivity to any of the components of the investigational product AGS67E:

  * AGS67E
  * L-Histidine
  * α-trehalose dihydrate or
  * polysorbate 20
* History of thromboembolic events (e.g., deep vein thrombosis (DVT) or pulmonary embolism (PE)) ≤ 2 weeks before the first dose of study drug and/or clinical diffuse intravascular coagulation (DIC)
* Active infection requiring treatment ≤7 days before the first dose of study drug
* Condition or situation which may put the subject at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study
* Any medical, psychiatric, addictive or other disorder which compromises the ability of the subject to give written informed consent and/or to comply with procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of adverse events | up to 34 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Concentration at the end of infusion (CEOI) | Escalation: Days 1-4, 8, 15, 22, 43-46, 50, 64 for Cycles 1-4 and predose once every 3 weeks in subsequent cycles. Expansion: Days 1, 3, 8, 22, 43, 45, 64 in Cycles 1-4 and predose once every 3 weeks in subsequent Cycles up to an average of 4 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Maximum observed concentration (Cmax) | Escalation: Days 1-4, 8, 15, 22, 43-46, 50, 64 for Cycles 1-4 and predose once every 3 weeks in subsequent cycles. Expansion: Days 1, 3, 8, 22, 43, 45, 64 in Cycles 1-4 and predose once every 3 weeks in subsequent Cycles up to an average of 4 months
Pharmacokinetic parameter for Monomethyl Auristatin E (MMAE): Time to maximum concentration (Tmax) | Escalation: Days 1-4, 8, 15, 22, 43-46, 50, 64 for Cycles 1-4 and predose once every 3 weeks in subsequent cycles. Expansion: Days 1, 3, 8, 22, 43, 45, 64 in Cycles 1-4 and predose once every 3 weeks in subsequent Cycles up to an average of 4 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Partial area under the serum concentration-time curve after first dose and as appropriate (AUC0-21) | Escalation: Days 1-4, 8, 15, 22, 43-46, 50, 64 for Cycles 1-4 and predose once every 3 weeks in subsequent cycles. Expansion: Days 1, 3, 8, 22, 43, 45, 64 in Cycles 1-4 and predose once every 3 weeks in subsequent Cycles up to an average of 4 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Terminal or apparent terminal half-life (t1/2) | Escalation: Days 1-4, 8, 15, 22, 43-46, 50, 64 for Cycles 1-4 and predose once every 3 weeks in subsequent cycles. Expansion: Days 1, 3, 8, 22, 43, 45, 64 in Cycles 1-4 and predose once every 3 weeks in subsequent Cycles up to an average of 4 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Systemic clearance (CL) | Escalation: Days 1-4, 8, 15, 22, 43-46, 50, 64 for Cycles 1-4 and predose once every 3 weeks in subsequent cycles. Expansion: Days 1, 3, 8, 22, 43, 45, 64 in Cycles 1-4 and predose once every 3 weeks in subsequent Cycles up to an average of 4 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Volume of distribution at steady state (Vss) | Escalation: Days 1-4, 8, 15, 22, 43-46, 50, 64 for Cycles 1-4 and predose once every 3 weeks in subsequent cycles. Expansion: Days 1, 3, 8, 22, 43, 45, 64 in Cycles 1-4 and predose once every 3 weeks in subsequent Cycles up to an average of 4 months

SECONDARY OUTCOMES:
Incidence of Anti-Drug Antibody (ADA) formation to the fully human monoclonal antibody (AGS67C) and antibody-drug conjugate (AGS67E) | Up to 34 months
Incidence of tumor response | Up to 34 months
  Tumor response is defined as either a complete response (CR) or partial response (PR)
Objective response rate (ORR) | Up to 34 months
  ORR for a cohort is defined as the percentage of subjects who experience a best response of either complete response (CR) or partial response (PR) in that cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (5):
- United States (4):
  - Site US0006, Duarte, California
  - Site US0002, Stanford, California
  - Site US0004, Fairway, Kansas
  - Site US0001, New York, New York
- Site CA0005, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=382